CLINICAL TRIAL: NCT01877902
Title: STUDY OF USE OF PEMETREXED IN PATIENTS WITH NON-SMALL LUNG CANCER METASTATIC IN ANDALUSIAN PUBLIC HEALTH SYSTEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FPS-PEM-2013-06
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pemetrexed 500 mg/m 2

SUMMARY:
STUDY OF USE OF PEMETREXED IN PATIENTS WITH NON-SMALL LUNG CANCER METASTATIC IN ANDALUSIAN PUBLIC HEALTH SYSTEM

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Confirmed diagnosis of metastatic NSCLC
* Pemetrexed Starts 1st line (either induction or maintenance) in any of the following periods:
* January 1, 2010 to March 31, 2010
* October 1, 2011 to December 31, 2011

Exclusion Criteria:

* Patients receiving pemetrexed within a clinical trial protocol because it is an experimental environment that does not reflect clinical practice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It will be included all patients diagnosed CPNMm participating centers to initiate treatment with pemetrexed in 1st line (either induction or maintenance.
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Determine utilization profile (line treatment and scheme used) of pemetrexed in patients with non-small cell lung cancer metastatic (CPNMm) in Andalusia. | 12 months

SECONDARY OUTCOMES:
1) Determine the progression-free survival and overall survival 2) Evaluate the degree of adherence in prescribing pemetrexed patients with CPNMm in Andalusia approved indications, the recommendations of the Pharmacy and Therapeutics Committees and | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Javier Bautista Paloma, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (18):
- Spain (18):
  - Hospital La Línea, Algeciras, Cádiz
  - Hospital Punta de Europa, Algeciras, Cádiz
  - Hospital Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Costa del Sol, Marbella, Cádiz
  - Hospital de Puerto Real, Puerto Real, Cádiz
  - Hospital de Baza, Baza, Granada
  - Hospital Universitario Torrecardenas, Almería
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital San Cecilio, Granada
  - Hospital Santa Ana, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Regional de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville